CLINICAL TRIAL: NCT00200512
Title: A Prospective, Randomized, Placebo-Controlled, Crossover Study of the Safety and Effectiveness of Subcutaneous Injections of Apomorphine in the Treatment of "Off" Episodes in Patients With "On/Off" or "Wearing Off" Effects Associated With Late Stage Parkinson's Disease
Brief Title: Continued Efficacy of Apomorphine After Previous Exposure of at Least Three Months
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APO301
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2000-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

INTERVENTIONS:
Drug: apomorphine HCl injection

SUMMARY:
The objective of this study was to measure the continued efficacy of apomorphine after previous exposure of at least three months duration.

DETAILED DESCRIPTION:
This was a prospective, double-blind, randomized, placebo-controlled, crossover desigh, multicenter study of the safety and effectiveness of subcutaneous apomorphine treatment. Patients received both apomorphine and placebo, in a randomized double-blind fashion

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson's Disease and classified as stage II-IV of the Hoehn and Yahr scale for staging the severity of Parkinson's Disease
* Patients must have been on an optimally maximized oral therapy regimen including levodopa/decarboxylase inhibitors in either immediate or delayed release forms, plus at least one direct acting oral dopamine agonist for at least 30 days prior to randomization
* Patients must have been receiving apomorphine subcutaneous injections for rescue therapy for "Off" events for at least three months with an average dosing requirement of at least 2 doses per day over the week prior to enrollment with a dose of less than 11 mg

Exclusion Criteria:

* Patients under medical therapy for clinically significant psychoses or dementia not related to ingestion of antiparkinson medications. (Patients with hallucinations or other central adverse reactions associated solely with antiparkinson medications were not excluded.)
* Patients with a history of drug or alcohol dependency within one year prior to study enrollment
* Patients with unstable and clinically significant disease of cardiovascular (including orthostatic hypotension), hematologic (including Coombs' positive hemolytic anemia), hepatic, renal, metabolic, respiratory, gastrointestinal or endocrinological systems or neoplasm within the threemonths before the start of the study.
* Patients with a history of allergy or intolerance to morphine or its derivatives, sulfur, sulfur containing medication, sulfites, domperidone, trimethobenzamide or other anticholinergics.
* Patients treated with experimental agents (other than apomorphine intermittent subcutaneous injections) within 3 months before study entry, experimental agents were defined on the basis of the regulatory status in the country of patient observation, or with other disallowed medications
* Patients whose apomorphine regimen was characterized by continuous infusion or by administration methods other than intermittent subcutaneous injection.
* Patients who could not or would not sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 1999-09; Study Completion 1999-11

PRIMARY OUTCOMES:
UPDRS Motor Score 20 minutes after dosing

SECONDARY OUTCOMES:
Dyskinesia Rating Scale 10, 20 and 60 minutes after dosing
Time to onset of perceived relief
AUC for UPDRS Motor Scores at predose, 10, 20 and 60 minutes
Change in UPDRS Motor Scores at 10 and 60 minutes after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Will Sullivan, Study Director — Mylan Bertek Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Walton Centre for Neurology and Neurosurgery, Liverpool
  - The Morriston Hospital, Swansea